CLINICAL TRIAL: NCT05875025
Title: Open-label, Randomised, Controlled, 2-way Cross-over Study to Assess the Effect of Multiple Doses of the New HFA-152a Propellant Versus the Marketed HFA-134a Propellant on Mucociliary Clearance in Healthy Volunteers
Brief Title: Study to Assess the Effect of the New HFA-152a Propellant on Mucociliary Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLI-05993AB6-06
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Mucociliary Clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Propellant (Experimental): Placebo HFA-152a propellant
  Interventions: Other: Placebo formulated with HFA-152a propellant via pMDI
- Reference Propellant (Placebo Comparator): Placebo HFA-134a propellant
  Interventions: Other: Placebo formulated with HFA-134a propellant via pMDI

INTERVENTIONS:
Other: Placebo formulated with HFA-152a propellant via pMDI — 5 inhalations BID (morning and evening) for 8 consecutive days, starting from the morning of Day 1 until the morning of Day 8
  Arms: Test Propellant
Other: Placebo formulated with HFA-134a propellant via pMDI — 5 inhalations BID (morning and evening) for 8 consecutive days, starting from the morning of Day 1 until the morning of Day 8
  Arms: Reference Propellant

SUMMARY:
The primary objective of this study was to assess the effect of multiple doses of the HFA-152a propellant and the HFA-134a propellant on mucociliary clearance (MCC).

DETAILED DESCRIPTION:
This clinical trial was a Phase I, single-centre, multiple-dose, randomised, open-label, controlled, 2-way cross-over study to assess the effect on MCC of the new HFA-152a propellant (5 inhalations BID for 8 days) versus the marketed HFA-134a propellant (5 inhalations BID for 8 days) in adult healthy volunteers by measuring the clearance from the lungs of inhaled radioaerosol.

A total of 20 subjects were randomised into the study.

Standard safety assessments was conducted during the Study, including safety blood and urine laboratory tests, vital signs, physical examinations, ECGs, spirometry, and observations of any adverse events (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Healthy male and female subjects aged 18-55 years (inclusive);
3. Ability to understand the study procedures, the risks involved and ability to be trained to use the inhalers correctly;
4. Body Mass Index (BMI) between 18 and 30 kg/m2 (extremes inclusive);
5. Non-smokers or ex-smokers who smoked < 5 pack-years and stopped smoking > 5 years prior to screening;
6. Good physical and mental status at screening and before randomisation;
7. Vital signs within normal limits at screening; body temperature < 37.5°C;
8. 12-lead digitised electrocardiogram (ECG) in triplicate considered as normal at screening;
9. Lung function measurements within normal limits at screening;
10. Female subjects fulfilling one of the following criteria: Women of non-childbearing potential (WONCBP). Women of childbearing potential (WOCBP) with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method preferably with low user dependency, from the signature of the informed consent form (ICF) and until the follow-up call.
11. Male subjects fulfilling one of the following criteria: Fertile male subjects with a pregnant or non-pregnant WOCBP partner: they must be willing to use male condom, from the signature of the ICF until the follow-up call.

Exclusion Criteria:

1. Participation in another clinical study with an investigational drug in the 3 months or five half-lives of that investigational drug (whichever is longer) preceding the administration of the study treatment;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorders ;
3. Clinically relevant abnormal laboratory values at screening;
4. Subjects with history of breathing problems (i.e. history of asthma including childhood asthma);
5. Positive serology test for human immunodeficiency virus (HIV) 1 or HIV2 serology at screening;
6. Positive results from the hepatitis serology, indicating acute or chronic hepatitis B or hepatitis C at screening;
7. Blood donation or blood loss (≥ 450 mL) during the 2 months prior to screening or randomisation;
8. Positive urine test for cotinine at screening or prior to randomisation;
9. Documented history of alcohol abuse within 12 months prior to screening, an average weekly alcohol intake of greater than 14 units, or a positive alcohol breath test at screening or prior to randomisation;
10. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen evaluated at screening or prior to randomisation;
11. Intake of non-permitted concomitant medications in the predefined period prior to screening or prior to randomisation;
12. Presence of any current infection, or previous infection that resolved less than 1 week prior to screening or to randomisation;
13. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the study;
14. Documented coronavirus disease 2019 (COVID-19) diagnosis within the last 2 weeks, or associated complications/symptoms which have not resolved within 2 weeks prior to screening or prior to randomisation;
15. Heavy caffeine drinker;
16. For females only: pregnant or lactating women;
17. The use of any kind of smoking electronic devices (e.g. e-cigarettes), within 6 months before screening or prior to randomisation;
18. Subjects for whom participation in this study will exceed a total radiation exposure of 5 mSv in the last 12-month period or 10 mSv in the last 5-year period;
19. Subjects with a total dosimetry value (including history of exposure through occupation) which contraindicates their participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BDD Pharma - Bio-Imaging Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 20 healthy male and female subjects 18-55y (inclusive) were enrolled according to the inclusion and exclusion criteria. They were randomised, to one of the two sequences with Test ([T], HFA-152a propellant) or Reference ([R], HFA-134a propellant), i.e. T-R sequence or R-T sequence, with 10 subjects per sequence. All the randomised subjects completed the study.
Groups:
- HFA-152a Followed by HFA-134a: HFA-152a and HFA-134a propellant via pressurised metered-dose inhaler (pMDI):
  Placebo formulated with HFA-152a propellant via pMDI: 5 inhalations BID (morning and evening) for 8 consecutive days, starting from the morning of Day 1 until the morning of Day 8.
  In this study arm, HFA-152a was used during period 1 and HFA-134a was used during period 2.
- HFA-134a Followed by HFA-152a: HFA-134a and HFA-152a propellant via pressurised metered-dose inhaler (pMDI):
  Placebo formulated with HFA-134a propellant via pMDI: 5 inhalations BID (morning and evening) for 8 consecutive days, starting from the morning of Day 1 until the morning of Day 8.
  In this study arm, HFA-134a was used during period 1 and HFA-152a was used during period 2.
Period: Overall Study
Arm/Group | HFA-152a Followed by HFA-134a | HFA-134a Followed by HFA-152a
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HFA-152a Followed by HFA-134a | HFA-134a Followed by HFA-152a | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (8.6) | 34.4 (5.9) | 34.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 1 | 1 | 2
  Hispanic | 0 | 1 | 1
  White | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 10 | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.15 (2.63) | 24.84 (2.89) | 25.50 (2.77)
Smoking status at screening [Count of Participants; unit: Participants]
  Ex-smoker | 2 | 1 | 3
  Non-smoker | 8 | 9 | 17
Lung Function Parameter -- FEV1 (actual value) [Mean (Standard Deviation); unit: L] | 3.877 (0.741) | 3.974 (0.730) | 3.926 (0.718)
FEV1 % of predicted normal value [Mean (Standard Deviation); unit: percent of predicted] | 102.81 (9.38) | 102.60 (8.55) | 102.71 (8.74)
FVC actual value [Mean (Standard Deviation); unit: L] | 4.835 (0.953) | 4.963 (0.895) | 4.899 (0.902)
FEV1/FVC [Mean (Standard Deviation); unit: Ratio] | 0.803 (0.040) | 0.802 (0.037) | 0.803 (0.037)

OUTCOME MEASURES:

1. Primary Outcome: Mucociliary Clearance Rate -- Right Whole Lung -- Percent Particle Retention at 2 Hours (PPR2) on Day 8
Description: MCC rate was assessed by the percent particle retention at 2 hours (PPR2) after the inhalation of radiolabelled particles.
  Results are shown as adjusted mean (95% CI) for change from baseline in PPR2 (right whole lung) on Day 8, considering either HFA-152a and HFA-134a propellants.
  PPR2=Percent particle retention at 2 h after the inhalation of radiolabelled particles
Time Frame: 2 hours post inhalation of radiolabelled particles
Population: The ITT analysis set, defined as all subjects who were randomised and received at least one dose of study treatment (analysed as randomised), included 20 subjects.
Measure: Mean (95% Confidence Interval); unit: percent of particle retention
Arm/Group | Test Propellant | Reference Propellant
Number analyzed (Participants) | 20 | 20
percent of particle retention | 0.94 [-1.47 to 3.34] | -0.42 [-2.82 to 1.98]
Statistical Analysis 1: Comparison: Test Propellant vs Reference Propellant; Test type: Other; p = 0.442, ANCOVA; Analysis of covariance (ANCOVA) model, included treatment, subject, and period as fixed effects; PPR2 at baseline as a covariate; Adjusted mean difference = 1.36, 95% CI 2-sided [-2.28 to 4.99]

2. Primary Outcome: Mucociliary Clearance Rate -- Right Whole Lung -- Percent Particle Retention at 4 Hours (PPR4) on Day 8
Description: Mucociliary Clearance rate (MCC) rate, as assessed by the percent particle retention (PPR) (in right whole lung) at 4 h after the inhalation of radiolabelled particles (PPR4), on Day 8.
  Results are shown as adjusted mean (95% CI) for change from baseline in PPR4 (right whole lung) on Day 8, considering either HFA-152a and HFA-134a propellants.
  PPR4=Percent particle retention at 4 h after the inhalation of radiolabelled particles
Time Frame: 4 hours post inhalation of radiolabelled particles
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of particle retention
Arm/Group | Test Propellant | Reference Propellant
Number analyzed (Participants) | 20 | 20
percent of particle retention | -0.58 [-2.29 to 1.14] | -1.27 [-2.99 to 0.44]
Statistical Analysis 1: Comparison: Test Propellant vs Reference Propellant; Test type: Other; p = 0.553, ANCOVA; Analysis of covariance (ANCOVA) model, included treatment, subject, and period as fixed effects; PPR4 at baseline as a covariate; Adjusted mean difference = 0.70, 95% CI 2-sided [-1.73 to 3.12]

3. Other Pre Specified Outcome: Mucociliary Clearance -- AUC(0-4) -- Right Whole Lung Region
Description: The MCC variables AUC(0-4) was calculated for PPR parameter on the right whole lung region up to 4 h after inhalation of the radiotracer.
  Results are shown as change from baseline (Day -1) and Day 8, as mean and SD, in percent x hour.
  AUC(0-4)=Area under the tracheobronchial particle retention curve between 0 and 4 h.
Time Frame: Post inhalation of radiolabelled particles; baseline and 4 h after inhalation of the radiotracer on Day 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent x h
Arm/Group | Test Propellant | Reference Propellant
Number analyzed (Participants) | 20 | 20
Percent x h | 1.093 (5.345) | -1.961 (6.402)

ADVERSE EVENTS:
Time Frame: The recording of adverse events (AEs) was the period starting from the time of the Informed Consent signature (Visit 1, Day 2 to 21 before Treatment period 1 (Day-1)) and until the subject's study participation ended at either an Early termination visit or a Follow-up visit or call ( 7-10 days after last intake of study treatment).
Description: A follow-up call (or visit) had to be performed in case of early termination as well, if the early termination visit was performed less than 7 days after the intake of the last dose of the study treatment.
  Safety set was used for the evaluation of AEs. Safety set included all subjects who were randomised and received at least one dose of study drug (HFA-152a or HFA-134a).
Arm/Group | Test Propellant | Reference Propellant
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Propellant (N=20) | Reference Propellant (N=20)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Balance Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of this study may be published or presented at scientific meetings. If a publication is presented by the Investigator, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (2):
  • Study Protocol (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT05875025/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT05875025/SAP_001.pdf